CLINICAL TRIAL: NCT00501423
Title: Antiplatelet Drug Resistances and Ischemic Events
Acronym: ADRIE
Status: Completed | Type: Observational
Sponsor: Pierre Fontana (Other)
Collaborators: Beziers Hospital (Other); University Hospital, Montpellier (Other); Ministry of Health, France (Other Government); Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Pierre Fontana, PI, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 06-034; CPP SUDMED IV 051201
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Symptomatic Atherothrombosis
Keywords: antiplatelet drug; resistance; atherothrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The ADRIE study is an observational study on the clinical relevance of platelet reactivity in aspirin and clopidogrel treated cardiovascular patients.

DETAILED DESCRIPTION:
The ADRIE study is an observational study on the clinical relevance of platelet reactivity in aspirin and clopidogrel treated cardiovascular patients.

Main objective:

* to determine if platelet reactivity, assessed by specific and non-specific tests, is predictive of ischemic events during the 3-year follow-up.

Secondary objectives:

* primary outcome in each pre-specified sub-group : patients with coronary artery disease, ischemic stroke or peripheral arterial disease as main qualifying disease at entry,
* to determine if platelet reactivity, assessed by specific and non-specific tests, is predictive of bleeding events during the 3-year follow-up,
* to investigate potential determinants of platelet reactivity at entry in the study

ELIGIBILITY:
Inclusion Criteria:

* Documented symptomatic ischemic atherothrombotic disease treated by aspirin, clopidogrel or both.

Exclusion Criteria:

* Known platelet disorder
* Chronic treatment by antiplatelet drugs other than aspirin or clopidogrel.
* Chronic anticoagulant treatment
* Chronic non steroid anti inflammatory drug treatment
* Active cancer
* Ongoing aspirin or clopidogrel treatment taken for more than 5 years prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Documented symptomatic ischemic atherothrombotic disease
Sampling Method: Probability Sample
Enrollment: 771 (Actual)
Dates: Start 2006-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
MACE | prospective follow-up
  adjudicating committee

SECONDARY OUTCOMES:
MACE in pre-specified sub-groups | prospective follow-up
  patients with coronary artery disease, ischemic stroke or peripheral arterial disease as main qualifying disease at entry

OTHER OUTCOMES:
potential determinants of platelet reactivity | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fontana, MD PhD, Principal Investigator — University Hospitals Geneva, Switzerland; Jean-Luc Reny, MD PhD, Principal Investigator — Beziers Hospital, France
Locations (1):
- University Hospital Geneva; Beziers and Monpellier University Hospitals, France, Geneva - Beziers - Montpellier, France

REFERENCES:
- [Derived] Reny JL, Berdague P, Poncet A, Barazer I, Nolli S, Fabbro-Peray P, Schved JF, Bounameaux H, Mach F, de Moerloose P, Fontana P; Antiplatelet Drug Resistances and Ischemic Events (ADRIE) Study Group. Antiplatelet drug response status does not predict recurrent ischemic events in stable cardiovascular patients: results of the Antiplatelet Drug Resistances and Ischemic Events study. Circulation. 2012 Jun 26;125(25):3201-10. doi: 10.1161/CIRCULATIONAHA.111.085464. Epub 2012 May 21. PMID 22615340
- [Derived] Fontana P, James R, Barazer I, Berdague P, Schved JF, Rebsamen M, Vuilleumier N, Reny JL. Relationship between paraoxonase-1 activity, its Q192R genetic variant and clopidogrel responsiveness in the ADRIE study. J Thromb Haemost. 2011 Aug;9(8):1664-6. doi: 10.1111/j.1538-7836.2011.04409.x. No abstract available. PMID 21692977